CLINICAL TRIAL: NCT03248427
Title: CORALLEEN: A Phase 2 Clinical Trial of Multi-agent Chemotherapy or Letrozole Plus Ribociclib (LEE011) as Neoadjuvant Treatment for Postmenopausal Patients With Luminal B/HER2-negative Breast Cancer.
Brief Title: Neadjuvant Multi-agent Chemotherapy or Letrozole Plus Ribociclib in Luminal B/HER2-negative Breast Cancer.
Acronym: CORALLEEN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SOLTI Breast Cancer Research Group (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOLTI1402
Record Dates: First submitted 2017-07-03; First posted 2017-08-14 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Neoadjuvant; Luminal B tumors; Ribociclib
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Letrozole; Doxorubicin; Cyclophosphamide; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ribociclib + Letrozol (Experimental): Ribociclib: 600mg, 3-weeks-on/-week-off treatment Letrozole: 2.5mg daily; Six 28 days cycles
  Interventions: Drug: Ribociclib; Drug: Letrozole 2.5mg
- Chemotherapy (Other): Chemotherapy treatment will consist of four cycles of AC (doxorubicin 60 mg/m2 and cyclophosphamide 600 mg/m2 every 21 days) followed by weekly paclitaxel during 12 weeks.
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel

INTERVENTIONS:
Drug: Ribociclib — Ribociclib flat-fixed dose of 600 mg daily (three 200-mg capsules), days 1 to 21 of a 28-days cycle.
  Other Names: LEE011
  Arms: Ribociclib + Letrozol
Drug: Letrozole 2.5mg — Daily continuous
  Arms: Ribociclib + Letrozol
Drug: Doxorubicin — 60 mg/m2 as a continuous IV perfusion
  Arms: Chemotherapy
Drug: Cyclophosphamide — 600 MG/M2 in a 30 minutes IV infusion
  Arms: Chemotherapy
Drug: Paclitaxel — 80 mg/m2, in one hour IV infusion
  Arms: Chemotherapy

SUMMARY:
CORALLEEN is a two-arm, randomized, multicentric study in postmenopausal women with primary HR+/HER2 negative Luminal B breast cancer that will explore if the combination of ribociclib with letrozole offers clinical benefit at least comparable to that of standard chemotherapy.

DETAILED DESCRIPTION:
This is a parallel, two-arm, randomized 1:1, stratified by tumor size and nodal involvement, open-label, multicenter, exploratory study in postmenopausal women with primary operable HR+/HER2-negative Luminal B breast cancer according to PAM50 intrinsic subtype to evaluate the clinical benefit and biological effects of ribociclib combined with letrozole.

The primary trial objective is to evaluate the ability of each treatment strategy to provide ROR-low score at surgery.

Luminal B patients will be randomized 1:1 to either letrozole plus ribociclib or chemotherapy.Two weeks after the first administration of the assigned treatment, patients will undergo a biopsy to assess early biological response to treatment, at Ki67 protein and gene expression level. After finalization of the assigned neoadjuvant treatment, patients will undergo surgery.

The primary endpoint, Rate of ROR-low (at surgery) after neoadjuvant treatment, according to the Prosigna test will be centrally assessed.

Baseline, Day 15 and post-treatment (surgical) primary breast tumor tissue samples should be available for each patient for molecular characterization A post-surgery visit will be performed within 28 days (7 days) from surgery, and will mark the end of the study for that patient

ELIGIBILITY:
Inclusion Criteria

1. Signed Informed Consent Form prior to any study-specific procedure.
2. Female patients.
3. Post-menopausal status and age ≥18 years.
4. Histologically confirmed invasive breast carcinoma, with all the following characteristics:

   * Primary tumor ≥ 2cm in largest diameter as measured by breast MRI
   * Stage I to stage IIIA breast cancer
   * No evidence of distant metastasis (M0)
5. Breast cancer eligible for primary surgery.
6. Available pre-treatment FFPE core (Tru-cut) biopsy evaluable for PAM50 or possibility to obtain one. Minimal sample requirements are to have at least 2 tumor cylinders with a minimal tissue surface of 10 mm2 tissue, containing at least 10% tumor cells and having enough tissue to do at least 2 cuts of 10 micrometers each.
7. Luminal B subtype as per PAM50 analysis of pre-treatment sample.
8. ER-positive and/or PgR-positive and HER2-negative tumor by ASCO/CAP guidelines assessed locally.
9. In the case of a multifocal tumor (defined as the presence of two or more foci of cancer within the same breast quadrant), the largest lesion must be ≥ 2 cm and designated the "target" lesion for all subsequent tumor evaluations and HR+/HER2-negative status must be documented in all the tumor foci.
10. ECOG performance status of 0 or 1.
11. Adequate hematological, renal and hepatic function.
12. Ability and willingness to comply with study visits, treatment, testing and to comply with the protocol.

Exclusion criteria

1. Any prior treatment for primary invasive breast cancer.
2. Inoperable locally advanced or inflammatory (i.e., inoperable Stage III) breast cancer.
3. Metastatic (Stage IV) breast cancer.
4. Bilateral invasive breast cancer.
5. Multicentric breast cancer, defined as the presence of two or more foci of cancer in different quadrants of the same breast.
6. Patients who have undergone sentinel lymph node biopsy prior to study treatment.
7. Inability or unwillingness to swallow pills.
8. Malabsorption syndrome or other condition that would interfere with enteric absorption of study drugs.
9. Participation in a prior investigational study within 30 days prior to enrollment or within 5 half-lives of the investigational product, whichever is longer.
10. Patient with a Child-Pugh score B or C.
11. Patient has active cardiac disease or a history of cardiac dysfunction including any of the following:

    * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty or stenting) or symptomatic pericarditis within 12 months prior to screening.
    * History of documented congestive heart failure (New York Heart Association functional classification III-IV).
    * Documented cardiomyopathy.
    * Patient has a Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO).
    * Clinical significant cardiac arrhythmias (e.g. ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g. bifascicular block, Mobitz type II and third-degree AV block)
    * Long QT Syndrome or family history of idiopathic sudden death or congenital long QT syndrome.
    * On screening 12-lead ECG, any of the following cardiac parameters (defined as the mean of triplicate ECGs: bradycardia (resting heart rate < 50), tachycardia (resting heart rate > 90), PR interval > 220 msec, QRS interval >109 msec, or QTcF interval ≥450 msec (using Fridericia's correction).
12. Uncontrolled hypertension (Systolic blood pressure >160 mmHg or <90 mmHg and/or diastolic >100 mmHg).
13. Active infection requiring intravenous (IV) antibiotics.
14. Symptomatic hypercalcemia despite adequate management.
15. Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis.
16. Known human immunodeficiency virus (HIV) infection.
17. Any other diseases, active or uncontrolled pulmonary dysfunction, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, that may compromise compliance with the protocol, that may affect the interpretation of the results, or renders the patients at high risk from treatment complications.
18. Significant traumatic injury within 3 weeks prior to initiation of study treatment.
19. Major surgical procedure (not including minor procedures such as lymph node biopsy, tumor core biopsy, fine needle aspiration) within 4 weeks prior to initiation of study treatment or not fully recovered from any side effects of previous procedures.
20. Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
21. History of other malignancy within 5 years prior to screening, except for appropriately treated basal or squamous cell carcinoma, carcinoma in situ of the cervix, non-melanoma skin carcinoma, or Stage I uterine cancer.
22. Hormone replacement therapy stopped less than 2 weeks before treatment start.
23. Currently receiving or has received systemic corticosteroids until 2 weeks before treatment start or who have not fully recovered from side effects of such treatment. Following corticosteroid uses are permitted: single doses, topical applications (e.g. for rash), inhaled sprays (e.g. for obstructive airways diseases), eye drops or local injections (e.g. intra-articular)
24. Known hypersensitivity to any of the excipients of ribociclib, letrozole, doxorubicin, cyclophosphamide or paclitaxel.
25. Patients currently on following medications, which cannot be interrupted 7 days prior treatment start:

    * Any prohibited medication as per letrozole, doxorubicin, cyclophosphamide, or paclitaxel label.
    * Herbal preparations/medications, dietary supplements.
    * Medications that have a known risk to prolong the QT interval or cause Torsades de Pointe.
    * Medications with a narrow therapeutic window and predominantly metabolized through CYP3A4/5.
    * Strong inducers or inhibitors of CYP3A4/5, including grapefruit, grapefruit hybrids, pummelos, star-fruit and Seville oranges.
    * Warfarin or other coumarin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin or fondaparinux is allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
Rate of ROR-low according to the Prosigna test. | 24 weeks
  Rate of ROR-low after neoadjuvant treatment at surgery, according to the Prosigna test,as per central assessment

SECONDARY OUTCOMES:
Tumor Overall response rate (ORR) | 24 weeks
  Tumor overall objective response rate (ORR), defined as the sum of Partial Responses (PR) and Complete Responses (CR) according to RECIST v1.1, as per Investigator's assessments by breast MRI.
pCR in the breast and axillary lymph nodes | 24 weeks
  pCR is defined as the complete absence of invasive carcinoma in the breast and axillary lymph nodes on histological examination.
PEPI Score | 24 weeks
  Preoperative endocrine prognostic index (PEPI) score in the ribociclib plus letrozole treatment arm compared to historical values
Residual Cancer Burden (RCB) | 24 weeks
  Rate of residual cancer burden (RCB) score 0 or 1 (RCB0/1) after neoadjuvant treatment, according to the MD Anderson Cancer Center procedures, as per central assessment.
Rate of breast conserving surgery (BCS) | 24 weeks
  Rate of breast conserving surgery
Decrease in Ki67 in both treatment arms. | At baseline, in week 2, and pre-surgery
  Decrease in Ki67 in both treatment arms.
Incidence, duration and severity of Adverse Events (AEs) | Up to 24 weeks
  Incidence, duration and severity of Adverse Events (AEs) assessed by the NCI Common Terminology for Classification of Adverse Events (CTCAE) version 4.

CONTACTS AND LOCATIONS:
Overall Officials: Aleix Prat, PhD, Principal Investigator — H.Clinic de Barcelona/; Joaquin Gavilá, MD, Principal Investigator — Fundación Instituto Valenciano de Oncología
Locations (21):
- Spain (21):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General de Catalunya, Barcelona
  - Hospital Universitari Vall d' Hebron, Barcelona
  - Institut Català d'Oncologia l'Hospitalet, Barcelona
  - Consorcio Hospitalario Provincial de Castellón, Castelló
  - Hospital San Pedro de Alcántara, Cáceres
  - Fundació Privada Hospital Asil de Granollers, Granollers
  - Centro Integral Oncologico Clara Campal, Madrid
  - Centro Oncológico MD Anderson International España, Madrid
  - Hospital Quirón Madrid, Madrid
  - Hospital Rey Juan Carlos, Madrid
  - Hospital Universitario 12 de octubre, Madrid
  - Hospital Universitario Fundación de Alcorcón, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitari Son Espases, Palma
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Virgen del Rocío, Seville
  - Hospital Virgen Macarena, Seville
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari Arnau de Vilanova de València, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Villacampa G, Falato C, Pare L, Hernando C, Arumi M, Saura C, Gomez G, Munoz M, Gil-Gil M, Izarzugaza Y, Ferrer N, Najera-Zuloaga J, Montano A, Ciruelos E, Gonzalez-Santiago S, Villagrasa P, Gavila J, Prat A, Pascual T. Pre-operative ribociclib plus letrozole versus chemotherapy: Health-related quality of life outcomes from the SOLTI CORALLEEN trial. Eur J Cancer. 2022 Oct;174:232-242. doi: 10.1016/j.ejca.2022.07.028. Epub 2022 Sep 5. PMID 36067616
- [Derived] Prat A, Saura C, Pascual T, Hernando C, Munoz M, Pare L, Gonzalez Farre B, Fernandez PL, Galvan P, Chic N, Gonzalez Farre X, Oliveira M, Gil-Gil M, Arumi M, Ferrer N, Montano A, Izarzugaza Y, Llombart-Cussac A, Bratos R, Gonzalez Santiago S, Martinez E, Hoyos S, Rojas B, Virizuela JA, Ortega V, Lopez R, Celiz P, Ciruelos E, Villagrasa P, Gavila J. Ribociclib plus letrozole versus chemotherapy for postmenopausal women with hormone receptor-positive, HER2-negative, luminal B breast cancer (CORALLEEN): an open-label, multicentre, randomised, phase 2 trial. Lancet Oncol. 2020 Jan;21(1):33-43. doi: 10.1016/S1470-2045(19)30786-7. Epub 2019 Dec 11. PMID 31838010